CLINICAL TRIAL: NCT05679115
Title: Randomized Evaluation of the Lifestyle Tool in Individuals With Type 2 Diabetes
Brief Title: Evaluation of Lifestyle Tool in Type 2 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HealthDiabetes2
Record Dates: First submitted 2022-12-29; First posted 2023-01-10 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle intervention (Experimental): Participants get access to the tool and use it regularly
  Interventions: Behavioral: Lifestyle tool
- Controls on standard care (No Intervention): Participants who get randomized to control cannot access the tool.

INTERVENTIONS:
Behavioral: Lifestyle tool — Regular use of the digital Lifestyle tool
  Arms: Lifestyle intervention

SUMMARY:
The overall aim of the study is to observe the change of long-term metabolic control in patients with type 2 diabetes who have access to a digital intervention tool as compared with randomized controls during one year. The tool is based on self-affirmation theory and has large emphasis on self-reflection to enable sustainable lifestyle changes. .

DETAILED DESCRIPTION:
Type-2 diabetes afflicts more than 300 million people worldwide and poses a heavy burden on the healthcare systems everywhere. Recent guidelines from the American Diabetes Association and the European Association for the Study of Diabetes recommend enhanced focus on lifestyle management in addition to glucose-lowering drugs. Individual or group-based diabetes education programs can improve glucose control and quality-of-life, but they are resource-intense and long-term outcomes are variable. Moreover, less than one out of ten individuals with diabetes attend such programs because of practical, medical and financial hurdles to attend sessions.

Consequently, there is a large need for complementary lifestyle support that can meet individual preferences in content and timing and reach many patients at low cost. Digital tools have considerable potential for clinical utility, but there are several important knowledge gaps. First, data on long-term efficacy (>6 months) are scarce. Second, they are often combined with coaching or intensified healthcare contacts, making it difficult to specifically assess the effect of the digital component and apply the results to a broad range of settings with variations in structure and resources. Third, it is unclear how they affect concrete behaviours such as physical activity and physiological measures of insulin resistance and insulin secretion.

The investigators have developed a self-managed lifestyle tool that is based on a new approach combining health information with structured self-reflection to effectively promote behavioural change. The tool is digital, does not require additional healthcare resources and could be used for large numbers of patients in a scalable manner.

Study participants with type 2 diabetes will now be randomized to access the tool and the change of long-term blood glucose from baseline to end of follow-up will be compared with participants who are randomized to a control group without access to the tool.

Participants attend study visits every three months for blood sampling. Study personnel are instructed to remain neutral at blood sampling visits and not reinforce usage in order to assess the frequency of use and resultant outcomes that can be expected in real-life situations over extended time without the need for increased healthcare support. Technical problems are referred to a study coordinator, who also responded to requests to clarify content in a general manner without providing personal advice.

Study participants are managed by their ordinary healthcare providers throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes at or above 35 years of age
* HbA1C at 52 mmol/mol or above
* Diagnosis of diabetes mellitus was based on prior documentation or treatment with anti-hyperglycemic medication
* written informed consent.

Exclusion Criteria:

* type 1 diabetes, MODY or secondary diabetes
* conditions or treatments that in the judgement of the Investigator could affect the study evaluation
* connection with the study team, funders, authorities, universities or other public or private bodies in such a way that specific interests in the study outcomes could be suspected.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of long-term blood glucose concentration measured as glycated hemoglobin at 1 year | 1 year
  Intraindividual change of long-term blood glucose concentration measured as glycated hemoglobin (HbA1c) at 1 year relative to baseline compared between participants with access to the tool and on usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Rosengren, Professor, Principal Investigator — Region Skåne
Locations (1):
- Clinical Research Center, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results will be shared after deidentification.
Time Frame: Data will be available after publication.
Access Criteria: To researchers who provide a methodologically sound proposal in order to achieve the aims of that proposal. Proposals should be directed by email to livsstilsverktyget@gu.se